CLINICAL TRIAL: NCT07227636
Title: Phase II Study of Adjuvant Botensilimab in Combination With Balstilimab in Patients With Colorectal Cancer and Persistent Circulating Tumor DNA Following Surgery and Chemotherapy
Brief Title: A Study of Botensilimab and Balstilimab for Colorectal Cancer With ctDNA+ After Surgery and Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-132
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Rectal Cancer
Keywords: Persistent Circulating Tumor DNA; Botensilimab; Balstilimab; ctDNA; ctDNA+; immunotherapy; checkpoint inhibitor; dual checkpoint blockade; AGEN1181; AGEN2034; CTLA-4 inhibitor; PD-1 inhibitor
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — balstilimab

STUDY DESIGN:
Intervention Model Description: This is a 2-part, 2-cohort each, phase II study. Part 2 is randomized.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1a: Stage III MSS Colorectal Cancer (Botensilimab and Balstilimab) (Experimental): All patients will receive botensilimab IV on day 1 of the 42 day cycle for 4 doses, balstilimab IV on days 1, 15, and 29 of the 42 day cycle. Patient then continues balstilimab alone for an additional two cycles IV on days 1, 15, and 29 of the 42 day cycle.
  Interventions: Drug: Botensilimab; Drug: Balstilimab
- Cohort 1b: MSS CRLM (Botensilimab and Balstilimab) (Experimental): All patients will receive botensilimab IV on day 1 of the 42 day cycle for 4 doses, balstilimab IV on days 1, 15, and 29 of the 42 day cycle. Patient then continues balstilimab alone for an additional two cycles IV on days 1, 15, and 29 of the 42 day cycle.
  Interventions: Drug: Botensilimab; Drug: Balstilimab
- Cohort 2a: Stage 3 MSS Colorectal Cancer (Botensilimab and Balstilimab vs. Placebo) Randomized (Experimental): All patients will receive botensilimab IV on day 1 of the 42 day cycle for 4 doses, balstilimab IV on days 1, 15, and 29 of the 42 day cycle. Patient then continues balstilimab alone for an additional two cycles IV on days 1, 15, and 29 of the 42 day cycle OR Placebo
  Interventions: Drug: Botensilimab; Drug: Balstilimab; Other: Placebo
- Cohort 2b: MSS CRLM (Botensilimab and Balstilimab vs. Placebo) Randomized (Experimental): All patients will receive botensilimab IV on day 1 of the 42 day cycle for 4 doses, balstilimab IV on days 1, 15, and 29 of the 42 day cycle. Patient then continues balstilimab alone for an additional two cycles IV on days 1, 15, and 29 of the 42 day cycle OR Placebo
  Interventions: Drug: Botensilimab; Drug: Balstilimab; Other: Placebo

INTERVENTIONS:
Drug: Botensilimab — All patients will receive botensilimab IV on day 1 of the 42 day cycle for 4 doses
  Other Names: AGEN1181
Drug: Balstilimab — All patients will receive balstilimab IV on days 1, 15, and 29 of the 42 day cyclePatient then continues balstilimab alone for an additional two cycles IV on days 1, 15, and 29 of the 42 day cycle.
  Other Names: AGEN2034
Other: Placebo — Placebo
  Arms: Cohort 2a: Stage 3 MSS Colorectal Cancer (Botensilimab and Balstilimab vs. Placebo) Randomized; Cohort 2b: MSS CRLM (Botensilimab and Balstilimab vs. Placebo) Randomized

SUMMARY:
The researchers are doing this study to find out whether the combination of botensilimab and balstilimab (BOT/BAL), followed by balstilimab alone, is an effective treatment for people with microsatellite stable (MSS) colorectal cancer or colorectal liver metastases (CRLM) who have measurable residual disease (MRD) after standard treatment with surgery and chemotherapy or total neoadjuvant therapy (TNT).

DETAILED DESCRIPTION:
This is a 2-part, 2-cohort each. Part-1 will be a non-randomized study of 54 subjects to assess ctDNA clearance, including 2 cohorts. Cohort 1a includes 27 patients with stage III non-MSI-H/pMMR colorectal cancer following surgery and adjuvant chemotherapy or total neoadjuvant therapy (TNT), with persistent MRD. Cohort 1b includes 27 patients with non-MSI-H/pMMR CRLM following surgery and peri-operative chemotherapy, with persistent MRD.

Part-2 will be a randomized, placebo-controlled, double-blind study of 230 patients with non- MSI-H/pMMR CRC with MRD, to assess RFS. Cohort 2a includes 113 patients with stage III non-MSI-H/pMMR colorectal cancer following surgery and adjuvant chemotherapy or TNT with persistent MRD, randomized 2:1 to treatment versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative, is willing and able to provide written informed consent.
* Histologically- or cytologically- confirmed colorectal cancer.
* ≥ 18 years of age on day of signing informed consent.
* Consent for use of archival tissue and blood draws for research purposes.
* Performance status of ECOG 0 or 1.
* Known non-MSI-H/pMMR by IHC, PCR or NGS testing. MSKCC confirmation of non-MSI-H/pMMR status is not mandatory prior to enrollment and treatment on the study. For patients with outside testing, if sufficient tissue is available testing may be repeated at MSKCC and will not impact initial eligibility.
* Consent to undergo MSK IMPACT or NGS, if not previously done
* Disease specific criteria:

  1. Cohorts 1a and 2a: Undergone a complete surgical resection (R0) for stage III colon or rectal cancer, followed by adjuvant chemotherapy with FOLFOX or CAPEOX. Post-operative chemotherapy not required if received previous oxaliplatin-based therapy. Total Neoadjuvant Therapy for rectal cancer with complete clinical and radiographic response is allowed.
  2. Cohorts 1b and 2b: Undergone a complete surgical resection (R0) for liver metastasis (ablation or stereotactic body radiation therapy [SBRT], but not Y-90, is permitted) and completed standard peri-operative chemotherapy. Peri-operative chemotherapy not required if received previous oxaliplatin-based therapy. Prior floxuridine via Hepatic Arterial Infusion Pump is permitted. Completed definitive treatment for the primary tumor including (R0) resection, or Total Neoadjuvant Therapy for rectal cancer with complete clinical and radiographic response.
* Positive ctDNA following completion of appropriate standard of care therapy.
* Patients must sign informed consent within 6 weeks of positive ctDNA result. The 6 weeks is considered from the date that the ctDNA is resulted, and not the date it is drawn.

Adequate organ function, defined as:

1. Absolute Neutrophil Count ≥ 1,500/mm3.
2. Platelet count ≥ 75,000/mm3.
3. Hemoglobin ≥ 9.0 g/dL
4. Creatinine clearance (CrCl) ≥60 mL/min.
5. AST and ALT ≤ 2.5 × ULN
6. Bilirubin ≤ 1.5 × ULN or Direct bilirubin ≤ ULN

   * Subjects of childbearing potential (or with partners of childbearing potential) must use effective contraception for the course of the study starting with the screening visit through at least 5 months after the last dose of study treatment. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom).

Exclusion Criteria:

* Presence of metastatic or recurrent disease.
* Known DNA polymerase epsilon (POLE) or DNA polymerase delta (POLD) activating mutation.
* R1 (microscopic residual tumor) or R2 resection (macroscopic residual tumor at resection margin).
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

  1. Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., dexamethasone containing antiemetic regimen or steroids as CT scan contrast premedication) may be enrolled.
  2. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* Hypersensitivity to botensilimab or balstilimab or any of its excipients.
* Chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent

  a. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* History of, or any evidence of active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* Current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 90 days after the last dose of trial treatment.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 agent.
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years of the start of study treatment (i.e., with use of disease-modifying agents or immunosuppressive drugs). The following are exceptions:

  1. Subjects with vitiligo or alopecia
  2. Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
* Known active TB (Bacillus tuberculosis).
* Uncontrolled infection with human immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required
* Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Patients who are receiving or who have received anti-HBV therapy and have undetectable HBV DNA prior to study entry are eligible. Serological testing for HBV at screening is not required.
* Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Patients on or who have received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for HCV at screening is not required.
* Received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Rate of ctDNA clearance (Cohort 1a) | 6 months
  The 6 months ctDNA clearance will be estimated using the binomial distribution along with exact 95% confidence intervals separately in each cohort.
Rate of ctDNA clearance (Cohort 1b) | 6 months
  The 6 months ctDNA clearance will be estimated using the binomial distribution along with exact 95% confidence intervals separately in each cohort.
Recurrence-free survival (RFS) (Cohort 2a) | 1 year
Recurrence-free survival (RFS) (Cohort 2b) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neil Segal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/